CLINICAL TRIAL: NCT07209410
Title: Impact of Brimonidine Tartrate Ophthalmic 0.025% on Patients Using Netarsudil 0.02%/Latanoprost 0.005% to Treat Glaucoma
Brief Title: Evaluating Injection With the Use of Brimonidine Tartrate Ophthalmic 0.025% on Patients Using Netarsudil 0.02%/Latanoprost 0.005% to Treat Glaucoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insight Eyecare Specialties, Inc. dba Vision Source Eyecare, (Other)
Responsible Party: Principal Investigator, Crystal Remington, Optometrist, Insight Eyecare Specialties, Inc. dba Vision Source Eyecare,
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSE002
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; Hyperemia
MeSH Terms: conditions — Glaucoma; Hyperemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brimonidine Tartrate (Experimental): Patients experiencing hyperemia greater than grade 2 on Efron scale will receive brimonidine tartrate (Lumify). Photo documentation of hyperemia and patient satisfaction questionnaires will be administered.
  Interventions: Drug: Brimonidine Tartrate Ophthalmic 0.025%

INTERVENTIONS:
Drug: Brimonidine Tartrate Ophthalmic 0.025% — Lumify is an approved eye drop to minimize ocular hyperemia.

SUMMARY:
To evaluate the effect of brimonidine tartrate 0.025% on conjunctival hyperemia in patients treated with netarsudil 0.02%/latanoprost 0.005% mono-therapy for intraocular pressure lowering.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients 18-65 years old diagnosed with open-angle glaucoma or ocular hypertension.

  2. Currently on netarsudil 0.02%/latanoprost 0.005% monotherapy for a minimum of 2-6 weeks.

  3. Able to move from current topical glaucoma treatment to netarsudil 0.02%/latanoprost 0.005% for a minimum of 4 weeks or longer based on FDA recommended washout per drug classification prior to Visit 3.

  4. Experience conjunctival redness as graded on the Efron scale of at least grade 2 after minimum of 4 weeks on netarsudil 0.02%/latanoprost 0.005% mono-therapy or longer based on recommended washout per drug classification 4. Have a best corrected Visual Acuity by Snellen chart of 20/30 or better in study eye.

  5. Are willing and able to self-administer or have an able person available to assist with administration of study drug.

Willing and able to comply with study procedures and attend follow-up visits.

Exclusion Criteria:

1. Allergy or hypersensitivity to brimonidine or other components of brimonidine tartrate 0.025% or netarsudil 0.02%/latanoprost 0.005%.
2. Use of any other topical ocular medications.
3. Active ocular infection, inflammation unrelated to glaucoma therapy, uveitis, iritis or congenital aphakia.
4. Have pterygium/pinguecula, chemosis, episcleritis, scleritis (or any condition that may affect hyperemia grading) in the opinion of the investigator
5. Have moderate or severe dry eyes.
6. Pregnant, plan to become pregnant or breastfeeding.
7. Concurrent or past use in the last 90 days of vasoconstrictive ocular drops other than brimondine 0.025%
8. Have undergone previous incision IOP lowering surgeries.
9. Have undergone previous laser surgery for glaucoma (selective laser trabeculoplasty (SLT) or argon laser trabeculoplasty (ALT)), or microinvasive glaucoma surgery (MIGS) with 6 months of screening.
10. Have had intraocular or per-ocular surgery within the past 3 months.
11. Advanced glaucoma or c/d ratio greater than 0.8. Are non-responsive to topical treatment with netarsudil 0.02%/latanoprost 0.005%.
12. In the judgement of the investigator, have previous or currently active clinically significant systemic or ocular disease in either eye that could affect study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Effron Grading scale of ocular redness | 2 weeks
  Measuring Ocular Hyperemia and injection.
  This is measured on Scale 0-4 0- Normal
  1. Trace
  2. Mild
  3. Moderate
  4. Severe

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Source, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided